CLINICAL TRIAL: NCT07283965
Title: Zanubrutinib and Acalabrutinib Use and Risk of Atrial Fibrillation in Patients With Chronic B-cell Malignancies
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco111525
Record Dates: First submitted 2025-11-26; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic B-cell Malignancies; BTK Inhibitors; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — zanubrutinib; acalabrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Zanubrutinib: Adult patients with a chronic B-cell malignancy exposed to zanubrutinib
  Interventions: Drug: Zanubrutinib
- Acalabrutinib: Adult patients with a chronic B-cell malignancy exposed to acalabrutinib
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Adult patients with a chronic B-cell malignancy exposed to zanubrutinib
  Groups: Zanubrutinib
Drug: Acalabrutinib — Adult patients with a chronic B-cell malignancy exposed to acalabrutinib
  Groups: Acalabrutinib

SUMMARY:
Background. Zanubrutinib and acalabrutinib are both associated with an increased risk of atrial fibrillation (AF) but AF comparative risk between these 2 BTK inhibitors (BTKis) remains largely unknown.

Objectives. Our aim was to examine the risk of developing incident AF with zanubrutinib exposure compared with acalabrutinib exposure.

Methods. Using the TriNetX research network database, authors will conduct a retrospective cohort analysis of deidentified, aggregate adult patients with chronic B-cell malignancies and exposed to zanubrutinib or acalabrutinib. Patients will be divided into 2 groups based on zanubrutinib or acalabrutinib exposure. After propensity score matching (PSM), Cox proportional hazard models will be used to calculate the hazard ratios (HRs) and 95% confidence intervals (CIs) to compare the 2 matched groups. The appropriateness of the proportional hazard assumption will be examined and risk differences (RDs) will be used if appropriate. Results will summarized with the use of Kaplan-Meier survival curves.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* diagnose with chronic B-cell malignancies
* exposed to zanubrutinib or acalabrutinib

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients - diagnose with chronic B-cell malignancies expose to zanubrutinib or acalabrutinib in the TrinetX database
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Risk of incident atrial fibrillation in patients exposed to zanubrutinib compared with those exposed to acalabrutinib in the matched cohort. | from the introduction of the BTK inhibitor and up to 5 years

SECONDARY OUTCOMES:
Risk of all-cause mortality in patients exposed to zanubrutinib compared with those exposed to acalabrutinib in thematched cohort | from the introduction of the BTK inhibitor and up to 5 years
Risk of incident intra-cerebral hemorrhage in patients exposed to zanubrutinib compared with those exposed to acalabrutinib in the matched cohort | from the introduction of the BTK inhibitor and up to 5 years
Risk of incident major bleeding in patients exposed to zanubrutinib compared with those exposed to acalabrutinib in the matched cohort | from the introduction of the BTK inhibitor and up to 5 years
Risk of incident hypertension in patients exposed to zanubrutinib compared with those exposed to acalabrutinib in the matched cohort | from the introduction of the BTK inhibitor and up to 5 years
Risk of incident MACE (composite) in patients exposed to zanubrutinib compared with those exposed to acalabrutinib in the matched cohort | from the introduction of the BTK inhibitor and up to 5 years
Risk of incident ventricular tachycardia/ventricular fibrillation/cardiac arrest (composite) in patients exposed to zanubrutinib compared with those exposed to acalabrutinib in the matched cohort | from the introduction of the BTK inhibitor and up to 5 months

IPD SHARING:
Plan to Share IPD: No
Actually, data from TrinetX are only freely available for health care organizations participating to the health research network database.